CLINICAL TRIAL: NCT00760136
Title: The Role of Quadriceps Contraction in Patellar Repositioning-a Computed Tomography Study
Brief Title: The Role of Quadriceps Contraction in Patellar Repositioning - a Computed Tomography Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: ethics committee of National Taiwan University Hospital, National Taiwan University Hospital
Other Study IDs: 9461712133
Record Dates: First submitted 2007-04-10; First posted 2008-09-26 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2008-09

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: patellofemoral pain; quadriceps contraction
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Computed Tomography — CT imaging of bilateral knee

SUMMARY:
Background Previous studies have a great discrepancy concerning the effects of quadriceps contraction on patellar lateral displacement and tilt in patients with patellofemoral pain syndrome. This discrepancy may be caused by lack of information regarding to classifications of patellofemoral alignment under quadriceps relaxed. We hypothesized quadriceps contraction has different effects on each type of patellofemoral malalignment.

Methods The investigators expect to recruit 150 subjects with patellofemoral pain syndrome to participate in this study. All patients underwent computed tomography imaging of symptomatic knees, with and without quadriceps muscle contraction in 0°, 15° and 30° of knee flexion. Patellar lateral condyle index and patellar tilt angles of Sasaki and modified Fulkerson were measured to investigate the effect of quadriceps contraction on patellar repositioning.

DETAILED DESCRIPTION:
Background Previous studies have a great discrepancy concerning the effects of quadriceps contraction on patellar lateral displacement and tilt in patients with patellofemoral pain syndrome. This discrepancy may be caused by lack of information regarding to classifications of patellofemoral alignment under quadriceps relaxed. We hypothesized quadriceps contraction has different effects on each type of patellofemoral malalignment.

We expect to recruit 150 subjects with patellofemoral pain syndrome to participate in this study. All patients underwent computed tomography imaging of symptomatic knees, with and without quadriceps muscle contraction in 0°, 15° and 30° of knee flexion. Patellar lateral condyle index and patellar tilt angles of Sasaki and modified Fulkerson were measured to investigate the effect of quadriceps contraction on patellar repositioning.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for patients with PFPS were suffering from pain with at least two kinds of knee-flexing activities such as:

  * sitting
  * getting up from sitting
  * walking upstairs or downstairs
  * squatting
  * getting up from squatting
  * running
  * kneeling
  * jumping

Exclusion Criteria:

The exclusion criteria included:

* The presence of any major medical disease
* Rheumatoid arthritis, gouty arthritis
* Recent history (within 3 months) of knee surgery
* Image findings of osteoarthritis
* Any deformity of lower limbs

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with patellofemoral pain.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2006-08; Study Completion 2009-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mai-Hwa Jan, MS, Study Director — Graduate institute of physical therapy
Locations (1):
- Mei-Hwa Jan, Taipei, Taiwan